CLINICAL TRIAL: NCT03067116
Title: Posturography Changes During Pregnancy
Status: Completed | Type: Observational
Sponsor: Caps Research Network (Other)
Responsible Party: Sponsor
Other Study IDs: CI-IRB-20160524-01
Record Dates: First submitted 2017-02-17; First posted 2017-03-01 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Pregnant Women
Keywords: balance, postural; fall risk; anthropometrics; blood pressure; SpO2; heart rate; heart rate variability; stance width
MeSH Terms: interventions — Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects: Adult, healthy pregnant women undergoing Posturography Evaluation, Anthropometrics, Vitals and answering Health and daily activity questionnaires
  Interventions: Diagnostic Test: Posturography Evaluation; Diagnostic Test: Anthropometrics; Diagnostic Test: Vitals; Other: Health and daily activity questionnaires

INTERVENTIONS:
Diagnostic Test: Posturography Evaluation — Posturography testing using the modified Clinical Testing of Sensory Integration in Balance (mCTSIB) protocol: the subjects will be required to stand on a hard or compliant surface in a comfortable posture, with eyes open or closed
  Other Names: Balance Testing; CAPS® Testing
Diagnostic Test: Anthropometrics — measurement of height, minimum stance width (feet together or as close as they can be), circumference of the torso at the breast level, of the abdomen, of the hip, and of each thigh, and supine fundal height
Diagnostic Test: Vitals — measurement (bilateral and seated/standing if applicable) of temperature, respiration rate, heart rate, blood pressure, pulse oxygenation and heart rate variability
Other: Health and daily activity questionnaires — one time general health questionnaire as well as session questionnaires asking the subjects if they have fallen since their last testing session and how comfortable they are in doing daily activities

SUMMARY:
Determine balance changes during pregnancy

DETAILED DESCRIPTION:
The subjects will be tested at enrollment and during weeks 20, 24, 28, 32, 36, 40 of their pregnancy, as well every 4 weeks postpartum up to 6 months. The following protocol will be used:

1. Subjects will also be asked to answer a short health questionnaire.
2. The following data will be recorded each time: height, minimum stance width, circumference measurements of the chest, abdomen, hip and each thigh as well as a supine fundal height. A full body side-profile photo was also taken to determine the curvature of the spine.
3. A session questionnaire will be used to determine if the subject had fallen or noticed any changes in their daily activity.
4. In a seated position, the following measurements will be recorded: 1-minute heart rate variability (HRV) with paced breathing, temporal scan body temperature, respiration rate, heart rate, blood pressure and SpO2 (these last three will be measured bilaterally).
5. Subject will undergo posturography testing using the modified Clinical Testing of Sensory Integration in Balance (mCTSIB) protocol: four 30 s tests in the following conditions: eyes open on a rigid surface (NSEO), eyes closed on a rigid surface (NSEC), eyes open on a compliant surface (PSEO), and eyes closed on a compliant surface (PSEC).
6. At the end of the posturography testing, heart rate, blood pressure and SpO2 will be re-measured bilaterally in the standing and then seated positions, as will be the seated HRV.

ELIGIBILITY:
Inclusion Criteria:

* healthy women less than 20 weeks pregnant

Exclusion Criteria:

* women affected by any pathology and/or more than 20 weeks pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult, healthy pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Stability Score | From enrollment to 6 month post partum
  The Stability Score (calculated as percentage ratio of the actual sway and the theoretical limit of stability) will be used to investigate how balance changes during pregnancy and how it correlates to anthropometrics, vitals and questionnaires

SECONDARY OUTCOMES:
Center of Pressure (CoP) coordinates | From enrollment to 6 month post partum
  The CoP coordinates (standard posturography measurements) will be also used to investigate how balance changes during pregnancy and how it correlates to anthropometrics, vitals and questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Elena Oggero, PhD, Principal Investigator — Caps Research Network
Locations (1):
- Innova Brain Rehabilitation, Marietta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] C.C. Keiser, N.D. Keiser, G. Pagnacco, E. Oggero "REPEATED EVALUATIONS OF FALL RISK AND POSTUROGRAPHIC CHANGES DURING PREGNANCY AND POST-PARTUM: A FEASIBILITY STUDY", Biomedical Sciences Instrumentation, 2017, Vol. 53, pp 269-75.